CLINICAL TRIAL: NCT06479655
Title: Compare the Efficacy and Outcome Between Fentanyl and Morphine as Analgo-sedation in Mechanically Ventilated Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohd Zulfakar Mazlan, MBBS, Associate Prof Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/KK/24010062
Record Dates: First submitted 2024-06-14; First posted 2024-06-28 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Fentanyl; Morphine

STUDY DESIGN:
Intervention Model Description: Randomized control trial, two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl (Active Comparator): Intravenous fentanyl infusion 0.5 - 1 mcg/kg/hr
  Interventions: Drug: Fentanyl
- Morphine (Active Comparator): Intraveous morphine infusion 0.05 - 0.1 mg/kg/hr
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl — Intravenous fentanyl infusion with dilution of 10mcg/ml
  Arms: Fentanyl
Drug: Morphine — Intravenous morphine infusion with dilution 1mg/ml
  Arms: Morphine

SUMMARY:
The primary aim of this clinical trial is to compare the effectiveness of fentanyl vs morphine as analgosedation in mechanically ventilated adult patients in the ICU. This study also aims to compare the outcomes of patients between the two groups.

The main questions it aims to answer are :

1. Does propofol and fentanyl infusion as analgo-sedation achieve targeted sedation score at 12 and 24 hours compared to propofol and morphine infusion in mechanically ventilated adult patients in the intensive care unit (ICU)?
2. Is there a difference between the proportion of patients requiring rescue sedation dose between the fentanyl and morphine groups?

DETAILED DESCRIPTION:
Researchers will randomize patients into 2 groups (Fentanyl and Morphine) and will start study drug accordingly for sedation in ICU.Proportion of patients from each group achieving targeted sedation score at 12 and 24 hours following initiation of the drug and proportion of patients from each group requiring rescue sedation dose will be recorded and analyzed.

Furthemore duration of mechanical ventilation, length of ICU stay and 14 days mortality rate will recorded and compared between this 2 groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Patients who are expected by the ICU team to require invasive mechanical ventilation in ICU for at least more than 24 hours and for whom the ICU team decides to initiate continuous infusion of sedation
* A patient who was ventilated and sedated not more than 12 hours before ICU admission.

Exclusion Criteria:

* Patients with chronic use of narcotics
* Patients with chronic liver failure or end-stage renal failure
* Patients with severe chronic neurocognitive dysfunction
* Patients with drug overdose
* Patients with a known allergy to either morphine or fentanyl
* Patients who are receiving neuromuscular blockers
* Patients who are pregnant
* Patients who are diagnosed to have severe traumatic brain in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
RASS score at 12 and 24 hours | 24 hours from study drug initiation
  To determine the proportion of patients achieving the targeted sedation guided by RASS score at 12 and 24 hours in both fentanyl and morphine group.
Rescue sedation doses | 24 hours from study drug initiation
  To determine the proportion of patients requiring rescue sedation doses between fentanyl and morphine group

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 90 Days
  To compare the duration of mechanical ventilation between the fentanyl and morphine groups
Length of ICU stay | 90 days
  To compare the length of ICU stay between the fentanyl and morphine groups
14 days mortality rate | 14 days from randomization
  To compare 14-day mortality rates between the fentanyl and morphine groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No